CLINICAL TRIAL: NCT04132063
Title: Efficacy and Safety of Generic Substitution of Original Levetiracetam in Patients With Epilepsy
Brief Title: Generic Substitution of Original Levetiracetam in Thai Epilepsy Patients
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/PY119
Record Dates: First submitted 2019-10-15; First posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Epilepsy
Keywords: Epilepsy; Generic; Levetiracetam; Therapeutic equivalency
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Generic levetiracetam
  Interventions: Drug: Generic levetiracetam

INTERVENTIONS:
Drug: Generic levetiracetam — Generic levetiracetam tablet as the same dose as original levetiracetam tablet at the switching date

SUMMARY:
The retrospective pre-post observational study was conducted to evaluate the real-world evidence of efficacy and tolerability of generic levetiracetam (oral tablet) which was switched from original levetiracetam (oral tablet) in patients with epilepsy at the national hospital for neurology and neurosurgery in Thailand. Epilepsy patients who received generic substitution to original levetiracetam at the same dose and had stable conditions of seizure were only included. In the period of 6 months, the investigators assessed the change of seizure frequency, the incidence of hospitalization due to breakthrough seizure, the incidence of adverse events and the incidence of composite outcomes related to dosage adjustment of antiepileptic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of epilepsy for at least 6 months prior to generic levetiracetam substitution;
* Same dosage form and strength of generic substitution to original levetiracetam;
* Stable dose of original levetiracetam and stable seizure frequency prior to generic levetiracetam substitution;
* Stable dose of generic levetiracetam after generic levetiracetam substitution

Exclusion Criteria:

* Absence seizure with levetiracetam monotherapy;
* Original levetiracetam in dosage form of oral solution or intravenous solution prior to generic levetiracetam substitution;
* Poor compliance;
* Death or loss of follow up;
* Unavailable data for evaluation of outcomes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any epileptic patients who received generic substitution to original levetiracetam from February 2016 to May 2018
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline seizure frequency | At baseline, 3 and 6 months after generic levetiracetam substitution
  Change from baseline seizure frequency per month at 3 and 6 months

SECONDARY OUTCOMES:
Hospitalization | During 6 months of generic levetiracetam substitution
  Incidence of hospitalization due to breakthrough seizure
Adverse events | During 6 months of generic levetiracetam substitution
  Incidence of adverse events after generic levetiracetam substitution
Composite outcomes | During 6 months of generic levetiracetam substitution
  Incidence of composite outcomes related to dosage adjustment of antiepileptic drugs such as
  1. Switching back to original levetiracetam due to experiencing an uncontrolled seizure or adverse drug reactions,
  2. The incremental dose of generic levetiracetam due to experiencing an uncontrolled seizure,
  3. The decremental dose of generic levetiracetam due to experiencing adverse events,
  4. Add-on other antiepileptic drugs due to experiencing an uncontrolled seizure,
  5. The incremental dose of concurrent antiepileptic drugs due to experiencing an uncontrolled seizure.

CONTACTS AND LOCATIONS:
Overall Officials: Jannapas Tharavichitkun, Principal Investigator — Mahidol University
Locations (1):
- Prasat Neurological Institute, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No